CLINICAL TRIAL: NCT02829359
Title: Effects of Antiviral Therapy on HBV Reactivation and Liver Function After Hepatectomy for HBV-DNA Negative HBV-related Hepatocellular Carcinoma
Brief Title: Effects of Antiviral Therapy on HBV Reactivation
Acronym: HBV-DNA(-)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Affiliated Tumor Hospital of Guangxi Medical University, Guangxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBV-DNA(-)/HCC
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2016-07

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entecavir therapy (Experimental): Patients who received entecavir (zhengda Tianqing Co., Ltd, Lianyungang, Jiangsu Province, China; 0.5 mg/d) were submitted to antiviral group. Patients in the antiviral group received entecavir begin in the first 3 days before surgery for at lest 1 month. No immunological therapy in perioperative period will be submitted to any included patients.
  Interventions: Drug: Entecavir therapy
- No antiviral therapy (No Intervention): Patients who did not receive any antiviral therapies were submitted as non-antiviral group. Patients in the non-antiviral group who underwent HBV reactivation will receive entecavir therapy. No immunological therapy in perioperative period will be submitted to any included patients.

INTERVENTIONS:
Drug: Entecavir therapy — Patients in the antiviral group received entecavir begin in the first 3 days before surgery for at lest 1 month.
  Arms: Entecavir therapy

SUMMARY:
Hepatitis B virus (HBV) reactivation happens after liver resection for HBV-related hepatocellular carcinoma (HCC) patients, particularly for those with positive serum HBV-DNA . The incidence rate and risk factors of HBV reactivation after hepatectomy for serum HBV-DNA negative HBV-related HCC are unclear.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) reactivation happens after liver resection for HBV-related hepatocellular carcinoma (HCC) patients, particularly for those with positive serum HBV-DNA . The incidence rate and risk factors of HBV reactivation after hepatectomy for serum HBV-DNA negative HBV-related HCC are unclear.From July 2012 to December 2015, 174 consecutive patients with serum HBV-DNA negative HBV-related HCC underwent resection were prospectively enrolled in the studied. There are 66 patients received preoperative antiviral therapy (antiviral group) and 108 patients did not receive any antiviral therapy (non-antiviral group). The incidence of HBV reactivation, risk factors of liver function were analyzed in perioperative period. HBV reactivation developed in 30 patients (27.8%) in the non- antiviral group and 2 patients (3.0%) in the antiviral group, respectively (P < 0.001). Multivariate analysis revealed that minor hepatectomy (HR, 4.695; 95% CI, 1.257-17.537, P = 0.021) and without antiviral therapy (HR, 8.164; 95% CI, 1.831-36.397, p =0.006) were risk factors attributed to HBV reactivation. Patients in antiviral group and non-antiviral group or reactivation group and without reactivation group have similar ALT, TBil, ALB, and PT in 7 days after resection. However, patients in antiviral group have significantly better ALT and ALB on day 30th after resection than those in control group. Moreover, similar phenomenon were observed when comparing those with or without HBV reactivation. Resection could lead to HBV reactivation during the perioperative period for serum HBV DNA negative HBV-related HCC, especially in patients who did not receive any antiviral therapy. Anti-HBV therapy can reduce the risk of reactivation, thus improving liver function after hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* underwent initial hepatectomy;
* preoperative serum HBsAg positive
* serum HBV DNA negative
* serum ALT in normal range
* Child-Pugh A liver function
* HCC was confirmed by histopathology
* patients in the treated group received Entecavir (ENT) while patients in the control group did not receive any antiviral therapy.

Exclusion Criteria:

* underwent preoperative TACE or other anti-tumor treatments
* underwent preoperative antiviral treatment for nearly a year
* with autoimmune disease, other organ malignant tumor, or other severe disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Rate of HBV reactivation | 1 month after surgery
HBV reactivation on the recovery of liver function | 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Le-Qun Li, MD, Study Director — Cancer Hospital of Guangxi Medical University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Li X, Zhong X, Chen ZH, Wang TT, Ma XK, Xing YF, Wu DH, Dong M, Chen J, Ruan DY, Lin ZX, Wen JY, Wei L, Wu XY, Lin Q. Efficacy of Prophylactic Entecavir for Hepatitis B Virus-Related Hepatocellular Carcinoma Receiving Transcatheter Arterial Chemoembolization. Asian Pac J Cancer Prev. 2015;16(18):8665-70. doi: 10.7314/apjcp.2015.16.18.8665. PMID 26745134
- [Background] Xie ZB, Zhu SL, Peng YC, Chen J, Wang XB, Ma L, Bai T, Xiang BD, Li LQ, Zhong JH. Postoperative hepatitis B virus reactivation and surgery-induced immunosuppression in patients with hepatitis B-related hepatocellular carcinoma. J Surg Oncol. 2015 Nov;112(6):634-42. doi: 10.1002/jso.24044. Epub 2015 Sep 30. PMID 26421419
- [Background] Jang JW, Kim YW, Lee SW, Kwon JH, Nam SW, Bae SH, Choi JY, Yoon SK, Chung KW. Reactivation of hepatitis B virus in HBsAg-negative patients with hepatocellular carcinoma. PLoS One. 2015 Apr 20;10(3):e0122041. doi: 10.1371/journal.pone.0122041. eCollection 2015. PMID 25894607
- [Background] Sohn W, Paik YH, Cho JY, Ahn JM, Choi GS, Kim JM, Kwon CH, Joh JW, Sinn DH, Gwak GY, Choi MS, Lee JH, Koh KC, Paik SW, Yoo BC. Influence of hepatitis B virus reactivation on the recurrence of HBV-related hepatocellular carcinoma after curative resection in patients with low viral load. J Viral Hepat. 2015 Jun;22(6):539-50. doi: 10.1111/jvh.12356. Epub 2014 Nov 7. PMID 25377516
- [Background] Lee JI, Kim JK, Chang HY, Lee JW, Kim JM, Chung HJ, Kim YS, Lee KS. Impact of postoperative hepatitis B virus reactivation in hepatocellular carcinoma patients who formerly had naturally suppressed virus. J Gastroenterol Hepatol. 2014 May;29(5):1019-27. doi: 10.1111/jgh.12472. PMID 24325315
- [Background] Huang L, Li J, Yan J, Sun J, Zhang X, Wu M, Yan Y. Antiviral therapy decreases viral reactivation in patients with hepatitis B virus-related hepatocellular carcinoma undergoing hepatectomy: a randomized controlled trial. J Viral Hepat. 2013 May;20(5):336-42. doi: 10.1111/jvh.12036. Epub 2012 Dec 5. PMID 23565616
- [Background] Lao XM, Luo G, Ye LT, Luo C, Shi M, Wang D, Guo R, Chen M, Li S, Lin X, Yuan Y. Effects of antiviral therapy on hepatitis B virus reactivation and liver function after resection or chemoembolization for hepatocellular carcinoma. Liver Int. 2013 Apr;33(4):595-604. doi: 10.1111/liv.12112. Epub 2013 Feb 13. PMID 23402625
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pubmed/28122361 — Oncotarget. 2017 Feb 28;8(9):15047-15056. doi: 10.18632/oncotarget.14789.